CLINICAL TRIAL: NCT00330083
Title: A RANDOMIZED, MULTIPLE DOSE, DOSE-ESCALATION, DOUBLE-BLIND, PLACEBO-CONTROLLED PHASE I TRIAL INVESTIGATING THE OPTIMAL SAFE DOSE OF ALK RAGWEED TABLET AMBROSIA ARTEMISIIFOLIA IN ADULT SUBJECTS WITH SEASONAL RHINOCONJUNCTIVITIS CAUSED BY RAGWEED POLLEN ALLERGY
Brief Title: Safety of ALK Ragweed Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RT-01
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: ALK Ragweed Tablet

SUMMARY:
This trial is performed to assess whether ALK Ragweed Tablet is safe to use in adults

ELIGIBILITY:
Inclusion Criteria:

* Ragweed pollen induced rhinoconjunctivitis
* Adults of either sex (18-50 years of age)
* Positive skin prick test to ragweed

Exclusion Criteria:

* Previous treatment with immunotherapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Assessment of safety by recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: George J. Atiee, MD, Principal Investigator — Healthcare Discoveries Inc.
Locations (1):
- Healthcare Discoveries Inc., San Antonio, Texas, United States

REFERENCES:
- [Derived] Christensen LH, Ipsen H, Nolte H, Maloney J, Nelson HS, Weber R, Lund K. Short ragweeds is highly cross-reactive with other ragweeds. Ann Allergy Asthma Immunol. 2015 Dec;115(6):490-495.e1. doi: 10.1016/j.anai.2015.09.016. Epub 2015 Oct 21. PMID 26507708